CLINICAL TRIAL: NCT06451237
Title: Weekend Systemic Isotretinoin for Maintaining Acne Remission: A Novel Approach
Brief Title: Acne Remission Maintenance by Weekend Systemic Isotretinoin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Carmen Ibrahim Farid, Professor of Dermatology, Venereology and Andrology, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0107396
Record Dates: First submitted 2024-05-01; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Intervention Model Description: Interventional study on 3 parallel groups, with random assignment and longitudinal follow up, conducted in two phases (treatment and maintenance).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessor responsible for the follow up (assessing primary and secondary measures) during the treatment and maintenance phases was blinded to the line of treatment used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Adapalene group (Active Comparator): Patients received full Isotretinoin course for treatment, and maintained on every other day adapalene gel.
  Interventions: Drug: Isotretinoin capsules
- Full Iso group (Active Comparator): Patients received full isotretinoin course for treatment, and maintained on weekend isotretinoin.
  Interventions: Drug: Isotretinoin capsules
- Clearance Iso (Active Comparator): Patients treated by systemic isotretinoin till full clearance and for a month thereafter, and maintained on weekend isotretinoin.
  Interventions: Drug: Isotretinoin capsules

INTERVENTIONS:
Drug: Isotretinoin capsules — A one year follow up for patients on three maintenance regimens after acne clearance, including weekend isotretinoin and adapalene gel.
  Other Names: Adapalene gel

SUMMARY:
The goal of this study is to learn if isotretinoin oral tablets as a weekend regimen are safe and effective to maintain freedom from acne lesions in young adults who have completed a full course of isotretinoin on daily basis and achieved total control of the acne activity.

DETAILED DESCRIPTION:
Three groups of adult acne patients will be given a full course of isotretinoin with a cumulative dose of 120-150 mg/Kg weight in the 1st two groups, and till lesional clearance in the 3rd group with an additional month of maintenance. Afterwards, the 1st group will use adapalene gel every other day for maintenance, the 2nd and 3rd groups will use weekend oral isotretinoin. Patients will be followed for a year for reappearance of acne lesions, and safety of maintenance regimens. Patients opinion will be also sought.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) with moderate to severe facial acne, as per the Investigator Global Assessment (IGA) scale

Exclusion Criteria:

* patients on systemic acne medications in the past 3 months or topicals in the last month, pregnant or breastfeeding females, those with evidence of endocrine disturbances or using medications for comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Incidence of acne relapse during maintenance phase | one year
  percent of patients having one grade worsening of their acne investigator global assessment scale achieved by end of treatment phase as assessed by the physician during follow up
Timing of acne relapse after initiating maintenance | one year
  The time interval between initiating maintenance and the occurrence of one grade worsening of the patient's investigator global assessment scale achieved by the end of treatment phase as assessed by the physician during follow up
Maximum severity of acne relapse during follow up | One year
  Maximum investigator global assessment score reached by the the patient during the follow up year
Incidence of adverse effects | One year
  Percent of patients reporting adverse effects in general, percent of patients reporting each category of side effects, including disturbed lipid profile, raised transaminases, psychological changes, dryness, hair shedding, ...

SECONDARY OUTCOMES:
subjective patient satisfaction by maintenance regimen | one year
  A patient oriented outcome, in which the patients are asked by the end of maintenance year to report their degree of satisfaction by the efficacy of maintenance regimen to prevent acne relapse on a visual analogue scale of 1-10, in which 1 is lowest satisfaction and 10 is highest satisfaction.
Subjective convenience of maintenance regimen to patient | one year
  A patient oriented outcome to assess the degree of convenience of the maintenance regimen for the patient as reported on a visual analogue scale of 1-10, where 1 is the lowest convenience, and 10 is the highest convenience.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Farid, MD, Principal Investigator — Professor of Dermatology
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No